CLINICAL TRIAL: NCT01620476
Title: A Randomised, Double-blind, Single-centre, Placebo-controlled, 21-day Multiple s.c. Doses, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Liraglutide (NNC 90-1170) in Healthy Japanese Male Subjects
Brief Title: Safety and Tolerability of Liraglutide in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1551
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 mcg/kg (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- 10 mcg/kg (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- 15 mcg/kg (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 5 mcg/kg for 21 days. Injected subcutaneously once daily. Progression to the next dose level based on safety data
  Arms: 5 mcg/kg
Drug: liraglutide — 5 mcg/kg for 7 days followed by 10 mcg/kg for 14 days. Injected subcutaneously once daily. Progression to the next dose level based on safety data
  Arms: 10 mcg/kg
Drug: liraglutide — 5 mcg/kg for 7 days followed by 10 mcg/kg for 7 days followed by 15 mcg/kg for 7 days. Injected subcutaneously once daily
  Arms: 15 mcg/kg
Drug: placebo — Liraglutide placebo administered to subjects randomised at each dose level in the ratio of 3:1

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to assess the safety and tolerability of liraglutide in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Japanese
* Body mass index (BMI) between 18 and 27 kg/m^2 inclusive

Exclusion Criteria:

* Any clinical laboratory values deviated from the reference range at the laboratory
* Presence of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders
* Hepatitis B surface antigen, Hepatitis C antibodies or HIV (human immunodeficiency virus) antibodies positive
* History of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders.
* History of significant allergy or hypersensitivity
* Known or suspected allergy to trial product or related products.
* History of drug or alcohol abuse
* Smokes more than 15 cigarettes, or the equivalent, per day andis unwilling to refrain from smoking whenever required for the trial procedure

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-09; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma liraglutide curve

SECONDARY OUTCOMES:
Cmax, maximum plasma liraglutide concentration
tmax, time to reach Cmax
Terminal phase elimination rate-constant
t½, terminal elimination half life
24-hour profiles of serum insulin
24-hour profiles of serum glucose
24-hour profiles of plasma glucagon
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Kageyama S, Hirao K, Shimizu A, Matsumura Y, Zdravkovic M, Rasmussen MF, Irie S. Tolerability, pharmacokinetics, and pharmacodynamics of liraglutide, long-acting human GLP-1 analogue - Phase 1 studies in Japanese healthy subjects with type 2 diabetes. Endocrinology and Diabetology 2007; 24 (6): 95-104
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com